CLINICAL TRIAL: NCT00824863
Title: An Open-Label, Proof of Concept Study to Determine the Safety and Efficacy of Ketoconazole 2% Foam in the Treatment of Pityrosporum Folliculitis
Brief Title: Safety and Efficacy of Ketoconazole 2% Foam in the Treatment of Pityrosporum Folliculitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wayne Fujita, M.D. (Individual)
Responsible Party: Sponsor-Investigator, Wayne Fujita, M.D., Principal Investigator, Fujita, Wayne, M.D.
Organization: Fujita, Wayne, M.D. (Individual)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U0275-502
Record Dates: First submitted 2009-01-15; First posted 2009-01-19 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Pityrosporum Folliculitis
Keywords: pityrosporum folliculitis; ketoconazole 2% foam
MeSH Terms: interventions — Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- one arm (Experimental): All 10 patients receive ketoconazole 2% foam in the uncontrolled study.
  Interventions: Drug: ketoconazole 2% foam

INTERVENTIONS:
Drug: ketoconazole 2% foam — topical antifungal foam to be applied to the folliculitis BID for 2-4 weeks.
  Other Names: ketaconozole 2% foam brand name is Extina Foam.

SUMMARY:
Pityrosporum folliculitis presents as fine superficial follicular pustules and papules on the trunk and upper extremities. Ketoconazole 2% foam was recently approved for the treatment of seborrheic dermatitis in immunocompetent patients 12 years and older. Ketoconazole 2% foam is felt to work by reducing the number of pityrosporum yeast organisms. Safety and efficacy of ketoconazole 2% foam treatment for this fungal infections has not been established. This study is to demonstrate efficacy and safety in the treatment of pityrosporum folliculitis.

DETAILED DESCRIPTION:
Malassezia/pityrosporum species is a ubiquitous saprophyte of human skin. This organism is implicated in the etiology of seborrheic dermatitis, tinea versicolor, and pityrosporum folliculitis. The prevalence of pityrosporum folliculitis is especially high in warm and humid environments, although its presence is universal. Pityrosporum folliculitis presents in immuno-competent, acne-prone young adults as fine superficial follicular pustules and papules on the trunk and upper extremities. There are no comedones. This acneiform condition is non-scarring. It causes significant morbidity for patients as it is frequently mistaken for acne vulgaris with scarring potential, often associated with pruritis, and fails to respond to adequate conventional acne treatment- systemic antibiotics, topical benzoyl peroxide, and topical retinoids. Pityrosporum folliculitis can be the sole presenting condition or it can coexist with acne vulgaris. Less commonly, patients with pityrosporum folliculitis present with associated tinea versicolor and seborrheic dermatitis. The diagnosis is made by clinical presentation, microscopic examination for the pustule for spores/hyphae, skin biopsy, and retrospectively following good response to antimycotic therapy.

Ketoconazole 2% foam was recently approved for the treatment of seborrheic dermatitis in immunocompetent patients 12 years and older. Safety and efficacy of ketoconazole 2% foam treatment for pityrosporum folliculitis has not been established. Prior to the availability of the ketoconazole 2% foam, successful treatment of pityrosporum folliculitis required systemic anti fungal drugs such as ketoconazole, itraconazole and fluconazole. It also responds to oral isotretinoin. Systemic antimycotics are effective but repeated use of these drugs incurs safety concerns including hepatotoxicity and drug-drug interactions. Oral isotretinoin is indicated for severe nodulo-cystic acne and generally is inappropriate as a routine treatment modality for pityrosporum folliculitis. As pityrosporum folliculitis is a non-scarring acneiform condition and can be recurrent, effective and safe, patient initiated topical treatment would be a more appropriate form of therapy.The objective of this study is to demonstrate that ketoconazole 2% foam may be the treatment of choice for pityrosporum folliculitis.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of pityrosporum folliculitis will be established by clinical presentation - fine, superficial follicular papules and pustules on the chest, back, and upper arms. KOH will be done on the pustules looking for spores and hyphae.
2. Concomitant acne treatments with standard acne treatment modalities will be allowed - oral and topical antibiotics, topical retinoids, and benzoyl peroxides.

Exclusion Criteria:

1. Pregnancy and breast feeding
2. Patients with nodulocystic acne on the trunk
3. Current or prior treatment with oral isotretinoin
4. Patients allergic to the ketoconazole topical foam product
5. Patients with associated serious systemic diseases or immunocompromised patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-12; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Lesion count reduction | 90 days

SECONDARY OUTCOMES:
Patient will be questioned on global assessment regarding response to treatment. | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Wayne H. Fujita, M.D., Principal Investigator — Private Practice
Locations (1):
- Aiea Medical Building; Suite 401, ‘Aiea, Hawaii, United States